CLINICAL TRIAL: NCT04977921
Title: An Authentic Solution to Translate Lab Skills Nursing Education Into Effective Clinical Practice During COVID-19: Elsevier Clinical Skill Platform
Brief Title: Lab Skills Nursing Education Into Effective Clinical Practice During COVID-19: Elsevier Clinical Skill Platform
Acronym: EDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Magda Bayoumi, Lecturer, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KKU2341751442
Record Dates: First submitted 2021-07-17; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Educational Problems
Keywords: Clinical lab session; Elsiever clinical skill; traditional lab session; students satisfaction

STUDY DESIGN:
Intervention Model Description: A quasi-experimental, two groups, pre-posttest study was carried out in Nursing college, King Khalid University, Kingdome of Saudi Arabia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elsiever clinical skill platform (Experimental)
  Interventions: Other: lab session

INTERVENTIONS:
Other: lab session — assign students to clinical modules for study the clinical lab scope of practice

SUMMARY:
This study aimed to investigate the effectiveness of utilizing an Elsevier clinical skill platform in clinical nursing education.

1.2. Research hypotheses

1. Nursing students who assign for the critical care clinical course modules using Elsevier clinical skill platform obtain a higher score in the OSCE than who receive clinical Lab session on campus.
2. Nursing students who utilize an Elsevier clinical skill are more satisfied in the clinical education journey.

DETAILED DESCRIPTION:
A quasi-experimental, two groups, pre-posttest study was carried out in Nursing college, King Khalid University, Kingdome of Saudi Arabia.

2.2 Instruments

1. Pre-posttest per skill was conducted for both group the Elsevier clinical skill group (ECS Group) and traditional Clinical Lab Session group (CLS Group), to assess the students' knowledge level before and after receiving each scheduled Lab Module.
2. Objective Structured Clinical Evaluation (OSCE): The summative OSCE included practical stations with an associated written paper for each skill examined. For the practical station, Students must pass the practical station (100%), as well as the relevant written station (70%) to achieve a pass in that scope of practice skill according to Exam policy & Procedure.
3. Students' perception of Usability and Learning of Elsevier Clinical Skill: included 8 questions developed by Rowe et al, 2017 categorized into two main themes: 1st theme is relevant to the Usability of the platform (4 items) and 2nd theme reflected the Learning enhancement while using the platform (4 items). Each item was scored on a three-point Likert scale as follows: Strongly agree or agree (3), Neither agree nor disagree (2) and Strongly disagree or disagree (1). The overall perceptions of students with both online and traditional lab experiences included and score ranged between (1-3) as 1= Much better than or better than, 2= About the same as 2, Much worse than or not as good as 3

2.3 Participants: A convenience sample of all students enrolled in the critical care nursing course (n=52) were divided into two groups and random selection was implemented by the registration office following the inclusion criteria for all students who were enrolled first time receive critical care nursing course. Therefore, two students were withdrawn at the beginning of the course. The first group represented the control group the Clinical Lab session (25 students), whilst the second group represented the intervention group the Elsevier clinical skill (25 students).

ELIGIBILITY:
Inclusion Criteria:

* Must be passed all prerequisite nursing courses

Exclusion Criteria:

* Unwilling to participate
* Request to use traditional lab session

Ages: 20 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Improve student's performance per clinical lab session | 13 lab session-13 weeks
  1. Pre-posttest per skill was conducted for both group the Elsevier clinical skill group (ECS Group) and traditional Clinical Lab Session group (CLS Group), to assess the students' knowledge level before and after receiving each scheduled Lab Module.
evaluate effectiveness of teaching pedagogy | Week 14
  2. Objective Structured Clinical Evaluation (OSCE): The summative OSCE included practical stations with an associated written paper for each skill examined. For the practical station, Students must pass the practical station (100%), as well as the relevant written station (70%) to achieve a pass in that scope of practice skill according to Exam policy & Procedure.

SECONDARY OUTCOMES:
assess students' perception of Usability and Learning of Elsevier Clinical Skill: | up to 15 weeks
  Included 8 questions 1st theme is relevant to the Usability of the platform (4 items) and 2nd theme reflected the Learning enhancement while using the platform (4 items). Each item was scored on a three-point Likert scale as follows: Strongly agree or agree (3), Neither agree nor disagree (2) and strongly disagree or disagree (1). The overall perceptions of students with both online and traditional lab experiences included and score ranged between (1-3) as 1= Much better than or better than, 2= About the same as 2, Much worse than or not as good as 3

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing Faculty, Abhā, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
data analysis completed July writing paper on August publish paper on September